CLINICAL TRIAL: NCT03406065
Title: The Effect of Sodium Bicarbonate Supplementation on Physical and Specific Performance Capacity in Combat Sports Athletes
Brief Title: Sodium Bicarbonate Supplementation in Combat Sports Athletes
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Poznan University of Life Sciences (Other)
Collaborators: Poznan University of PhysED (Individual)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: ULS00003
Record Dates: First submitted 2018-01-14; First posted 2018-01-23 (Actual); Last update posted 2018-01-23 (Actual); Status verified 2018-01

CONDITIONS: Supplementation; Sport
Keywords: Sodium bicarbonate; NaHCO3; Combat Sports; Physical capacity; Dummy test

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sodium bicarbonate supplementation (Experimental): Group taking oral NaHCO3 supplementation in a progressive-dose regimen.
  Interventions: Dietary Supplement: Sodium bicarbonate supplementation
- Placebo treatment (Placebo Comparator): Group taking oral supplementation with placebo (maltodextrin with NaCl) in a similar tablet form prepared by the same producer as NaHCO3 tablets.
  Interventions: Dietary Supplement: Placebo treatment

INTERVENTIONS:
Dietary Supplement: Sodium bicarbonate supplementation — The experimental procedure for each athlete included a 10-day NaHCO3 supplementation in a progressive-dose regimen in order to reduce the likelihood of gastrointestinal side effects (from 25 to 100 mg ∙ kg-1). NaHCO3 was administered in the form of unmarked disk-shaped tablets (Alkala T, SANUM, Poland). The tablets were ingested with at least 250 mL of water and could be either swallowed or dissolved in the mouth. On training days the supplements were taken in the morning, in the evening and 1.5 hours before training session. On rest days the supplements were taken in the morning, in the afternoon and in the evening.
  Arms: Sodium bicarbonate supplementation
Dietary Supplement: Placebo treatment — The experimental procedure for each athlete included a 10-day placebo administration. Placebo was ingested with at least 250 mL of water. On training days the supplements were taken in the morning, in the evening and 1.5 hours before training session. On rest days the supplements were taken in the morning, in the afternoon and in the evening.
  Arms: Placebo treatment

SUMMARY:
The purpose of this study was to verify the effect of 10-day sodium bicarbonate (NaHCO3) and placebo (PLA) supplementation on physical and specific performance capacity, as well as concentrations of the selected biochemical blood markers in trained combat sports athletes, in a randomised, double-blind, placebo-controlled trial.

DETAILED DESCRIPTION:
Sodium bicarbonate (NaHCO3) was proposed as an ergogenic agent, because it improves high-intensity and resistance exercise performance. Until now the major limitation to NaHCO3 supplementation has been the gastrointestinal (GI) side effects. Therefore, this study aims to examine the effect of chronic, progressive-dose NaHCO3 ingestion on physical capacity and specific performance capacity, and concentrations of the selected biochemical blood markers in trained combat sports athletes, in a randomised, double-blind, placebo-controlled trial.

ELIGIBILITY:
Inclusion Criteria:

* written informed consent from all participants before the study (included aslo informed consents to the participation in the study of athletes under the age of 18 obtained from their parents)
* a current medical clearance to practice sports,
* training experience: at least 4 years (of combat sport training),
* minimum of 4 workout sessions (combat sport) a week,

Exclusion Criteria:

* current injury,
* any health-related contraindication,
* declared general feeling of being unwell,
* unwilling to follow the study protocol.

Ages: 17 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 64 (Actual)
Dates: Start 2014-10-10 (Actual); Primary Completion 2015-01-20 (Actual); Study Completion 2015-04-05 (Actual)

PRIMARY OUTCOMES:
Changes in anaerobic capacity after sodium bicarbonate supplementation | Baseline and after 10 days
  The Wingate Anaerobic Test (WAnT)
Changes in specific performance capacity after sodium bicarbonate supplementation | Baseline and after 10 days
  The wrestler's special endurance test - projective test with dummy (DT)

SECONDARY OUTCOMES:
Changes of lactate and pyruvate concentration in blood after sodium bicarbonate supplementation | Baseline and after 10 days
  Lactate [mmol/L] and pyruvate [mmol/L] concentration analysis
Changes of creatine kinase and lactate dehydrogenase activity in blood after sodium bicarbonate supplementation | Baseline and after 10 days
  Creatine kinase [U/L] and lactate dehydrogenase [U/L] activity analysis
Changes in blood glucose and hemoglobin concentration after sodium bicarbonate supplementation | Baseline and after 10 days
  Hemoglobin (Hb) [g/dl] and glucose [g/dl] concentration analysis
Changes in blood hematocrit levels after sodium bicarbonate supplementation | Baseline and after 10 days
  Hematocrit (HCT) [%] level analysis
Changes of red and white blood cell concentration in blood after sodium bicarbonate supplementation | Baseline and after 10 days
  Red blood cells (RBC) [mln/mm³] and white blood cells (WBC) [mln/mm³] concentration analysis
Changes in polyphenols and albumin concentration | Baseline and after 10 days
  Polyphenols [g/L] and and albumin [g/L] concentration analysis
Changes in FRAP concentration | Baseline and after 10 days
  FRAP [µmol/L] concentration analysis

CONTACTS AND LOCATIONS:
Overall Officials: Jan Jeszka, Professor, Study Chair — Poznan University of Life Sciences, ul. Wojska Polskiego 31, Poznań, Wielkopolska, Poland, 60-624
Locations (1):
- Poznan University of Life Sciences, ul.Wojska Polskiego 31, Poznan, Wielkopolska, Poland

IPD SHARING:
Plan to Share IPD: Undecided
Shared data will be exclusively related to the level recorded indicators (anaerobic capacity and specific performance capacity indicators, levels of biochemical markers, body composition), without personal data. The data obtained will be attached to scientific publications, depending on the requirements of the journal.